CLINICAL TRIAL: NCT04341480
Title: The Safety of Chemotherapy for Patients With Gynecological Malignancy in High-risk Region of COVID-19, a Prospective Cohort Study
Brief Title: The Safety of Chemotherapy for Patients With Gynecological Malignancy in High-risk Region of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: 2020-TJ-COVID-19
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Gynecological Cancer
Keywords: COVID-19; SARS-CoV-2; Gynecological cancer; Chemotherapy
MeSH Terms: conditions — COVID-19 | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy group: Routine chemotherapy every 3 weeks for 2 cycles, and follow up for 2 weeks after discharge from hospital. Total observation duration is 6 weeks.
  Interventions: Drug: Chemotherapy
- Control group: No treatment, based on patient's choice. Total observation duration is 6 weeks.

INTERVENTIONS:
Drug: Chemotherapy — Routine chemotherapy for individual tumor type.
  Groups: Chemotherapy group

SUMMARY:
A novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) disease (COVID-19) emerged at December 2019 in Wuhan, China, and soon caused a large global outbreak. The delayed treatment for many chronic diseases, due to the concern of SARS-CoV-2 infection, is an increasing serious problem. Here the investigators investigate the safety of chemotherapy for patients with gynecological malignancy in Wuhan, the center of high-risk regions of COVID-19.

DETAILED DESCRIPTION:
A novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; previously provisionally named 2019 novel coronavirus or 2019-nCoV) disease (COVID-19) emerged at December 2019 in Wuhan, Hubei Province, China. This infectious disease soon caused a large global outbreak and became a major public health issue. As of 19:00, 12 March 2020, the total number of confirmed cases of SARS-CoV-2 in China has reached 80982 with 3173 death, and 110 other countries have officially reported 45164 cases of SARS-CoV-2 infection with 1520 death.

In this particular time, only patients with SARS-CoV-2 or other diseases with an emergency condition were receipted by most of the hospitals in Hubei Province, even in many other regions of China. The delayed treatment for many chronic diseases, such as malignant tumors, is an increasing serious problem. One major concern was that patients with malignant tumors were generally older in age with low immunity. Preliminary study has shown that cancer patients are most susceptible to infect SARS-CoV-2 and more likely to develop a severe pneumonia. But many other researches suspected that conclusion. Moreover, many of the patients with malignant tumors are facing short term death from tumors rather than the risk of infection. Nevertheless, there is not sufficient evidence to insure the safety of chemotherapy in high-risk region of COVID-19, and there is also not sufficient information to judge which patients' tumor therapy can be appropriately delayed. Here the investigators investigate the safety of chemotherapy for patients with gynecological malignancy in Wuhan, the center of high-risk regions of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 80 years old female.
* Patient must have histologically confirmed either type of gynecological malignancies.
* Chemotherapy must be essential for the patient.

Exclusion Criteria:

* Diagnosed or suspected patients with covid-19 pneumonia, according to the symptom, nucleic acid tests, antibody tests for SARS-CoV-2, or CT scan of the lungs.
* Patient has a prior SARS-CoV-2 infection without clinical cure for 28 days.
* Patient has close contact with diagnosed or suspected SARS-CoV-2 infected person within 14 days.
* Patient has inadequate general condition, severe complication or organ dysfunction not fit for chemotherapy (based on the judgment of researchers).
* Patient or the family refuses to sign the informed consent.
* Patient does not cooperate in following up.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecological malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | through study completion, an average of 3 months.
  Incidence rate of SARS-CoV-2 infection within the whole period of the study.

SECONDARY OUTCOMES:
Tumor response | 6 weeks after enrollment.
  Tumor response by determining changes (PD, SD, PR, CR) according to Response Evaluation Criteria in Solid Tumours (RECIST), version 1.1
Safety and tolerability of chemotherapy as measured by the Common Terminology | through study completion, an average of 3 months.
  Safety and tolerability of chemotherapy as measured by the Common Terminology Criteria for Adverse Events (version 4.0)
Quality of Life (QOL) measures using Functional Assessment of Cancer Therapy (FACT- ovarian cancer) | through study completion, an average of 3 months.
  To evaluate quality of life (QOL) for the subjects undergoing this treatment, using validated tools. QOL will be assessed every 3 months during treatment course. [Functional Assessment of Cancer Therapy - Ovarian Cancer questionnaire (score range from 0 to 160. Higher scores represent better quality of life.
  questionnaire core-30 (QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided